CLINICAL TRIAL: NCT00744133
Title: An Interventional Plasmodium Falciparum Malaria Challenge Model Utilizing the NF54 Strain of Parasite Transmitted by Aseptic A. Stephensi Mosquitoes to Healthy Malaria-Naïve Adult Volunteers
Brief Title: Malaria Challenge With NF54 Strain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 05-0053; Malaria CVD 17000; N01AI80057C
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-07

CONDITIONS: Plasmodium Falciparum Infection
Keywords: Plasmodium falciparum, NF54, Anopheles stephensi, mosquito, malaria
MeSH Terms: conditions — Malaria, Falciparum; Malaria

ARMS (2):
- Group 1: 1, 3, or 5 bites (Experimental): Part A: 18 subjects receive 1, 3, or 5 bites of Anopheles stephensi mosquitoes infected with the NF54 strain of Plasmodium falciparum.
  Interventions: Biological: NF54 P. falciparum isolate
- Group 2: N bites (Experimental): Part B: 20 subjects receive N bites of Anopheles stephensi mosquitoes infected with the NF54 strain of Plasmodium falciparum.
  Interventions: Biological: NF54 P. falciparum isolate

INTERVENTIONS:
Biological: NF54 P. falciparum isolate — 1, 3, 5 or N bites from aseptically-raised Anopheles stephensi female mosquitoes infected with Plasmodium falciparum parasites of the NF54 strain.

SUMMARY:
The purpose of this study is to determine how many infected mosquito bites are required to reliably give volunteers a case of malaria. It is expected that volunteers will develop malaria and may have symptoms. Safety is the main concern. A malaria challenge is given by allowing a volunteer to receive 1, 3, or 5 mosquito's bites. Then participants are carefully followed and blood is tested. The study will also look at how immune systems (the cells and substances that protect the body from infection and foreign matter) respond after mosquito bite challenges. About 38 subjects (aged 18-40 years) from the greater Baltimore, Maryland (United States) community will participate and may stay overnight for 10 days at a local medical center. Procedures include medical screening, assignment to a dose group, a mosquito bite challenge, and 56 day follow-up. Volunteers will be contacted by telephone at 6 and 12 months after the malaria challenge.

DETAILED DESCRIPTION:
This is a randomized trial of the aseptically raised anopheles mosquito malaria challenge. Adults aged 18-40 years will be randomized to one group of 18 subjects (Part A) or a second group of 20 subjects (Part B). Adults will be randomized to receive 1, 3 or 5 bites of Anopheles (A.) stephensi mosquitoes infected with the NF54 strain of chloroquine-sensitive Plasmodium (P.) falciparum. Part B will be informed by the results of Part A. Thus, a total of approximately 38 adults will receive a malaria challenge. The challenge for Part A will be given on day 0 with the subsequent group (Part B) commencing after a 56 day safety review. Solicited adverse events will be recorded on the days of malaria challenge, outpatient days 5-7, 19-28, 35, 42, 49, and 56 post-challenge event. Inpatient analysis will occur from Days 8-18 or until three-day directly observed therapy for P. falciparum infection is complete. Additional outpatient, post-malaria infection follow-up will occur weekly for 4 weeks. Unsolicited adverse events will be recorded for 56 days after each malaria challenge event. Participants will receive a telephone follow-up six and twelve months after enrollment. The primary objective is to develop and evaluate the safety and tolerability of a new human malaria challenge model using aseptically-raised anopheles mosquitoes infected with the NF54 isolate of P. falciparum and reared under current Good Manufacturing Practices (cGMPs) conditions. Secondary objectives are to obtain information on the minimum number of A. stephensi bites required to safely achieve 100 percent adult human volunteer infectivity (Malaria challenge, Part A); obtain information on the minimum quantity of A. stephensi bites in a second challenge study to achieve 100 percent adult human volunteer infectivity (Malaria challenge, Part B); develop molecular diagnostic techniques for rapid and accurate real-time diagnosis of P. falciparum infection to assess the role as a new diagnostic standard for P. falciparum challenge studies.

ELIGIBILITY:
Inclusion Criteria:

* Male or nonpregnant female between the ages of 18 and 40 years, inclusive.
* Women who are not surgically sterile (no history of bilateral tubal ligation, bilateral salpingo-oophorectomy, or hysterectomy), post-menopausal (1 year without menses) or determined otherwise by medical evaluation to be sterile must agree to practice adequate contraception [such as double barrier methods (condoms plus foam or spermicide, diaphragm plus foam or spermicide), some intrauterine devices (IUDs), intravaginal or transdermal hormonal methods initiated at least 1 month prior to inoculation, or a vasectomized partner] for the entire study period (56 days). Serologic pregnancy tests will be conducted upon screening. Urine testing will be done on the day of malaria challenge, on the day of the first positive malaria smear and at the conclusion of active surveillance (Day 56).
* Is in good health, as determined by vital signs (heart rate, blood pressure, oral temperature), medical history, screening 12-lead electrocardiogram (ECG) and a physical examination.
* Has normal laboratory values [urinalysis (assessing blood and protein presence as greater than trace by dipstick), hemoglobin, white blood cells, platelet count, aspartate aminotransferase (AST), (alanine aminotransferase) ALT, glucose and creatinine] prior to challenge study.
* Able to understand and comply with planned study procedures including an inpatient stay from Day 8-18 after malaria challenge.
* Provides informed consent prior to any study procedures, correctly answers greater than or equal to 70 percent on the post consent quiz and is available for all study visits.
* Willing to avoid non-study related blood donation for 3 years following Plasmodium falciparum challenge.

Exclusion Criteria:

* Has any known history of malaria infection, is a long-term resident (> 5 years) of a malaria-endemic area, was born and resided in a malaria-endemic area, or has traveled to a malaria-endemic area within the previous 6 months.
* Has a positive urine pregnancy test prior to malaria challenge (if female of childbearing potential), is lactating, or has the intention to become pregnant within 2 months after enrollment in this study.
* Use of any antibiotic or antimalarial drug beginning 28 days prior to the screening and extending to Day 56 of study surveillance.
* Has evidence of increased cardiovascular disease risk (defined as > 10 percent, 5 year risk) as determined by the method of Gaziano. Risk factors include sex, age (years), systolic blood pressure (mm Hg), smoking status (current versus past or never), body mass index (BMI) (kg/mm^2), reported diabetes status (yes/no), current treatment for raised blood pressure (yes/no).
* Is immunosuppressed (e.g., poorly-controlled diabetes mellitus, cirrhosis, renal insufficiency, active malignancy, connective tissue disease, organ transplant) as a result of an underlying illness or treatment.
* An abnormal electrocardiogram (EKG), defined as one showing pathologic Q waves and significant ST-T wave changes; left ventricular hypertrophy; any non-sinus rhythm excluding isolated premature atrial contractions; right or left bundle branch block; or advanced (secondary or tertiary) A-V heart block.
* Has an active neoplastic disease (excluding nonmelanotic skin cancer) or neoplastic disease within the past 5 years or any history of hematologic malignancy.
* Is using or intends to continue using oral or parenteral steroids, high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs (an exception includes asthma for which any oral or inhaled steroid intake will mean exclusion from study enrollment).
* Has a known active history of human immunodeficiency virus, hepatitis B surface antigen positivity, or hepatitis C infection.
* Has a history of active alcohol or drug abuse in the last 5 years.
* Has a history of receiving blood products within the 3 months prior to enrollment in this study.
* Has a history of psoriasis or porphyria, which may be exacerbated after treatment with chloroquine.
* Has an acute or chronic medical condition that, in the opinion of the investigator, would render malaria challenge unsafe or would interfere with the evaluation of responses (this includes, but is not limited to: known liver disease, renal disease, neurological disorders, visual field defects, cardiac disorders, pulmonary disorders, auditory damage, diabetes mellitus, and transplant recipients).
* Has a history of anaphylactic response to mosquito bites or known allergy to chloroquine, 4-aminoquinoline derivatives [atovaquone/proguanil (Malarone®)], ibuprofen, or acetaminophen that may be used to treat volunteers developing malaria after Plasmodium falciparum challenge.
* Is using or intends to continuing using a medication known to cause drug reactions with chloroquine or Malarone®, such as cimetidine, metoclopramide, antacids or kaolin (antacids and kaolin can be administered at least 4 hours from intake of chloroquine).
* History of retinal or visual field changes, auditory damage, or seizures.
* History of splenectomy.
* Has known sickle cell trait or laboratory evidence of sickle cell trait.
* Has an acute illness, including an oral temperature greater than 100.4 degrees Fahrenheit, within 1 week prior to malaria challenge.
* Plans to undergo surgery (elective or otherwise) between enrollment and 4 weeks (28 days) post-challenge.
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to enrollment in this study, or expects to receive an experimental agent during the 2-month post-challenge period.
* Has a diagnosis of schizophrenia, bi-polar disease or other major psychiatric disease.
* Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Occurrence of a positive malaria smear after the malaria challenge. | During a 56-day surveillance period (day of challenge and days 5-28, 35, 42, 49, and 56 after challenge).
Occurrence of serious adverse events. | After malaria challenge during a 56-day surveillance period (day of challenge and days 5-28, 35, 42, 49, and 56 after challenge) and 10 month follow-up period
Occurrence and severity of solicited symptoms. | 7 days after the malaria challenge and for the duration of follow-up after a malaria event (treatment days x 3 and smear-negative x 2 plus weekly follow-up x 4).
Occurrence and severity of unsolicited adverse events. | After malaria challenge during a 56-day surveillance period (day of challenge and 55 subsequent days. Volunteers will be questioned at Visits 2-29).

SECONDARY OUTCOMES:
Occurrence of a positive real-time quantitative polymerase chain reaction (PCR). | After malaria challenge during a 56-day surveillance period (day of challenge and days 5-28, 35, 42, 49 and 56 after challenge).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Background] Laurens MB, Billingsley P, Richman A, Eappen AG, Adams M, Li T, Chakravarty S, Gunasekera A, Jacob CG, Sim BK, Edelman R, Plowe CV, Hoffman SL, Lyke KE. Successful human infection with P. falciparum using three aseptic Anopheles stephensi mosquitoes: a new model for controlled human malaria infection. PLoS One. 2013 Jul 16;8(7):e68969. doi: 10.1371/journal.pone.0068969. Print 2013. PMID 23874828
- [Background] Lyke KE, Laurens M, Adams M, Billingsley PF, Richman A, Loyevsky M, Chakravarty S, Plowe CV, Sim BK, Edelman R, Hoffman SL. Plasmodium falciparum malaria challenge by the bite of aseptic Anopheles stephensi mosquitoes: results of a randomized infectivity trial. PLoS One. 2010 Oct 21;5(10):e13490. doi: 10.1371/journal.pone.0013490. PMID 21042404